CLINICAL TRIAL: NCT03891563
Title: Prospective Evaluation of Sport Activity and the Development of Femoroacetabular Impingement in the Adolescent Hip (PREVIEW)
Brief Title: Prospective Evaluation of Sport Activity and the Development of Femoroacetabular Impingement in the Adolescent Hip
Acronym: PREVIEW
Status: Active, not recruiting | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: McMaster Surgical Association (Unknown); Arthroscopy Association of North America (Other); Conmed (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: PREVIEW
Record Dates: First submitted 2019-03-25; First posted 2019-03-27 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2024-11

CONDITIONS: Femoroacetabular Impingement
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sport specialists, MVPA: AOSSM Criteria:
  1. Participation in intensive training and/or competition in organized sports greater than 8 months per year (essentially year round)
  2. Participation in 1 sport to the exclusion of participation in other sports (limited free play overall)
  3. Involving prepubertal (seventh grade or roughly age 12 years) children.
  AND
  Activity Tracker Criteria:
  Greater than 180 accumulated minutes of moderate-to-vigorous physical activity (MVPA) during participation in one sport type across one week of activity tracking
  - Meets these criteria within either one or both years of follow-up
- Non-sport specialist, any activity level: AOSSM Criteria:
  1. Participation in more than 1 sport at any physical activity level OR
  2. Participation in none or low training and/or competition in organized sports for any period of time.
  3. Involving prepubertal children.
  AND
  Activity Tracker Criteria:
  Greater than or less than 180 accumulated minutes of MVPA across one week of activity tracking
  - Meets these criteria during both years of follow-up

SUMMARY:
Femoroacetabular impingement (FAI) is a condition of the hip where there is a mis-fit between the femoral head (ball) and hip acetabulum (socket). The abnormalities on the hip bones collide or "impinge" during movements such as hip flexion and rotation. Typically, patients with this condition are young adults who present with hip pain, loss of hip function, and in many cases, osteoarthritis later in life. The rate of diagnoses of FAI has dramatically risen across all age groups, but it has been especially notable within adolescent populations. There has been a corresponding increase in the number of surgeries performed on younger and younger hips to treat pain and loss of function due to this condition. Preliminary small-scale research has hypothesized that increased activity, such as sport specialization (i.e. playing only one sport for most of the year) at an early age when the hip is still developing, may be the cause. In the past 20 years, sport injuries among children have dramatically increased, where close to 45 million young athletes participate in organized sports annually in Canada and the US alone. There is a current trend among coaches and parents to have children focus on one sport with the thought that this dedication will allow them to reach an elite level. We are proposing the first international, longitudinal cohort study to determine the effect of sport specialization on the development of FAI during the critical phase of hip development (i.e. between the ages of 12-14 years). Volunteer participants will be recruited across Canada and internationally and will be evaluated clinically and radiographically (i.e. using MRI) over 2 years. This study will not only prospectively evaluate the role of sport activity the development of FAI, but also inform preventative training protocols to potentially reduce its incidence among adolescents, and later as adults, as well as identify parameters to detect hips that are at risk for developing FAI.

DETAILED DESCRIPTION:
This is a multi-centre, international longitudinal cohort study evaluating 200 participants between the ages of 12-14 that include sport specialists at the moderate to vigorous physical activity (MVPA) level and non-sport specialists at any activity level. Participant groups will be defined according to the AOSSM and AMSSM early sport specialization criteria (2016). We will monitor physical activity levels of all participants using an activity log and a wrist-mounted activity tracker, with synced data collected every 3 months during the study period. In addition, participants will be evaluated clinically and radiographically at time of enrollment and 6, 12, 18, and 24 months. The primary study outcome is the incidence of FAI between groups at 2 years, determined via MRI. Secondary outcomes include hip function and health-related quality of life between subjects diagnosed with FAI versus no FAI at 2 years, as determined by the HOS and PedsQL questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. asymptomatic males and females between the ages of 12-14 years
2. ability to speak, understand, and read the language of the clinical site
3. provision of informed child assent (if applicable) and parental consent.

Exclusion Criteria:

1. hip is mature (i.e. closed physes) based on the baseline MRI scan
2. hip complaints or pain in the hip
3. previous trauma to the hip
4. previous surgery on the hip
5. significant medical co-morbidities (requiring daily assistance for ADLs)
6. history of or ongoing paediatric hip disease (Legg-Calve-Perthes; slipped capital femoral epiphysis, hip dysplasia)
7. participants that have contraindications and/or are unwilling to undergo an MRI (e.g. claustrophobia)
8. participants who will likely have problems, in the judgment of the investigator, with maintaining follow-up
9. any other reasons the investigator feels is relevant for excluding the subject.

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population will be comprised of adolescents aged 12-14 with no prior or ongoing hip comorbidities, and consent to receiving MRI scans at baseline and 2 years.
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of radiographic FAI | 2 years
  The primary outcome is the incidence of radiographic FAI between groups at 2 years, as determined by the dedicated MRI of the hip. We will identify both symptomatic and asymptomatic cases, where asymptomatic FAI can become symptomatic in young adulthood, and/or could be associated with idiopathic osteoarthritis later in life.

SECONDARY OUTCOMES:
Hip function | 2 years
  As determined by the Hip Outcome Score
Health-related quality of life | 2 years
  As determined by the Pediatric Quality of Life questionnaire

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (2):
  - McMaster University, Hamilton, Ontario
  - Chu du Quebec, Québec, Quebec
- Erasmus Medical Centre, Rotterdam, Netherlands
- Kyungpook National University Hospital, Daegu, Gyeongsangbuk-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ohlin A, Simunovic N, Duong A, Ayeni OR; PREVIEW investigators. Protocol for a multicenter prospective cohort study evaluating sport activity and development of femoroacetabular impingement in the adolescent hip. BMC Musculoskelet Disord. 2020 Apr 11;21(1):221. doi: 10.1186/s12891-020-03220-6. PMID 32278355